CLINICAL TRIAL: NCT05361408
Title: A Single Center, Open-label, Parallel, Phase IV Clinical Trial to Evaluate Efficacy of Once or Twice ZOledronic Acid After Different Duration of denOsumMab Administration in Postmenopausal Women With Osteoporosis
Brief Title: A Clinical Trial to Evaluate Efficacy of Once or Twice ZOledronic Acid After Different Duration of denOsumMab Administration in Postmenopausal Women With Osteoporosis (ZOOM Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1023
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab short-term user (Active Comparator): Denosumab injection less than 5 times
  Interventions: Drug: Zoledronic acid, once
- Denosumab long-term user (Active Comparator): Denosumab injection more than 5 times
  Interventions: Drug: Zoledronic acid, twice

INTERVENTIONS:
Drug: Zoledronic acid, once — Intravenous infusion of 5mg zoledronic acid, once
  Other Names: Zoledronate
  Arms: Denosumab short-term user
Drug: Zoledronic acid, twice — Intravenous infusion of 5mg zoledronic acid for 6month interval, twice
  Other Names: Zoledronate
  Arms: Denosumab long-term user

SUMMARY:
Denosumab(Dmab) is a monoclonal antibody that inhibits the receptor-activator of nuclear factor kappa-B ligand. It improves bone density and reduces fractures by inhibiting osteoclast recruitment and differentiation. Although the FREEDOM trial showed Dmab increase bone mineral density for ten years, the effect was reversible. When Dmab is discontinued, the rebound phenomenon, the bone mineral density returns to the pre-treatment value, and multiple vertebral fractures may occur. Recently, a guideline to administer bisphosphonates sequentially when Dmab is discontinued has been published. In several studies, Zoledronic acid prevented bone loss after denosumab discontinuation with a single administration in Dmab short-term(less than 2.5years) users, but in Dmab long-term(more than 2.5years) users, zoledronic acid did not fully prevent loss of BMD. Our study tried to evaluate that ZOL administration twice for six months apart in long-term Dmab users is not inferior to a single administration of ZOL in Dmab short-term users.

DETAILED DESCRIPTION:
Background Dmab is an osteoporosis treatment that improves bone density and lowers the risk of fractures. However, in a recent study, it is known that cases in which bone density decreases and multiple vertebral fractures occur when Dmab is discontinued. Therefore, the guideline recommends using zoledronic acid sequentially when discontinuing Dmab. However, the effect of preserving bone mineral density in patients who discontinue Dmab after using a long period is still not known.

Aim To investigate the difference in lumbar bone mineral density between the two groups when zoledronic acid was administered differently according to the administration period after discontinuation of denosumab in postmenopausal osteoporosis patients.

Methods A prospective, single-center, open-label, parallel, intervention study in 114 patients investigating the difference in bone mineral density between the short-term denosumab group and long-term denosumab group when zoledronic acid was administered differently. Each group is classified into a short-term group when used for less than 2.5 years and a long-term group when used for more than 2.5 years according to the maintenance period of the denosumab. The short-term group administrates zoledronic acid once six months after the last denosumab injection, and the long-term group administrates zoledronic acid six months and 12 months after the last denosumab injection, respectively. In the long-term group, if the side effect is severe after the first zoledronic acid administration and additional administration is difficult, it can be replaced with risedronic acid and maintained for another six months. The patients will be monitored with DXA at baseline and 12 months. Bone turnover marker (b-crosslap(CTx), P1NP) will be monitored at 6 and 12 months after the infusion of the first zoledronic acid. Whole spine x-rays are taken at baseline and 12 months after the zoledronic acid injection to check for vertebral fractures.

Perspectives Osteoporosis is a disease that requires continuous management in old age. In order to prevent fractures, the order and maintenance of drug administration should be decided from a long-term perspective. Denosumab is a potent inhibitor of bone resorption which can be used in patients with high risk and very high fracture risk. But since it is reversible, additional treatment must be continued to maintain bone mass when the drug is discontinued. This study will show if two injections of zoledronic acid six months apart in long-term denosumab patients can effectively prevent bone loss compared to a single administration of zoledronic acid in the short-term denosumab group.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (defined as no menstruation for more than 48 weeks prior to screening and no other pathological or physiological causes. If in doubt, a serum follicle-stimulating hormone (FSH) test may be performed at screening)
2. Patients diagnosed with osteoporosis, osteoporotic fractures, received at least two doses of denosumab, and who have osteopenia in follow-up DXA

Exclusion Criteria:

1. Secondary osteoporosis (Systemic glucocorticoid use, aromatase inhibitor, thyrotoxicosis, hypeparathyroidism, etc)
2. Active cancer treatment
3. Inflammatory bowel disease
4. History of medication related osteonecrosis of jaw(MRONJ)
5. low-energy fracture within the last 12months
6. Estimated glomerular filtration rate (eGFR) < 35 mL/min
7. Hepatic dysfunction (aspartate transaminase (AST)/alanine transferase (ALT) > 3 x upper normal limit)
8. Contraindication for zoledronic acid according to the SPC
9. Allergic to zoledronic acid

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 114 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
BMD lumbar spine | One year
  Change in lumbar spine BMD from baseline to one year after the zoledronic acid infusion

SECONDARY OUTCOMES:
BMD Femoral neck and total hip | One year
  Changes in femoral neck and total hip BMD from baseline to one year after the zoledronic acid infusion
Bone turnover marker | One year
  Changes in p-CTX and P1NP From Baseline to Six and twelve months After the Zoledronic Acid Infusion.
Vertebral fracture | One year
  Morphometric Vertebral Fractures Assessed by whole spine x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsourdi E, Zillikens MC, Meier C, Body JJ, Gonzalez Rodriguez E, Anastasilakis AD, Abrahamsen B, McCloskey E, Hofbauer LC, Guanabens N, Obermayer-Pietsch B, Ralston SH, Eastell R, Pepe J, Palermo A, Langdahl B. Fracture risk and management of discontinuation of denosumab therapy: a systematic review and position statement by ECTS. J Clin Endocrinol Metab. 2020 Oct 26:dgaa756. doi: 10.1210/clinem/dgaa756. Online ahead of print. PMID 33103722
- [Background] Solling AS, Harslof T, Langdahl B. Treatment With Zoledronate Subsequent to Denosumab in Osteoporosis: A 2-Year Randomized Study. J Bone Miner Res. 2021 Jul;36(7):1245-1254. doi: 10.1002/jbmr.4305. Epub 2021 Apr 20. PMID 33813753